CLINICAL TRIAL: NCT03476005
Title: Technology Enhanced Learning and Proficiency Based Progression to Investigate and Mitigate 'Wrong Blood in Tube' in Our Hospitals; Can we Improve Patient Safety and Reduce Resource Wastage?
Brief Title: Proficiency Based Training to Investigate WBIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Patrick Henn (Other)
Responsible Party: Sponsor-Investigator, Patrick Henn, Lecturer Medical Education, University College Cork
Organization: University College Cork (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: #1710
Record Dates: First submitted 2017-07-05; First posted 2018-03-23 (Actual); Last update posted 2018-07-05 (Actual); Status verified 2018-07

CONDITIONS: Transfusion Related Complication; Wrong Blood in Tube

STUDY DESIGN:
Intervention Model Description: Incidence of wrong blood in tube in interns provided with proficiency based progression training supported by technology enhanced learning in 2017 will be compared with historical controls from the same period in 2016
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Proficiently Trained interns - (Active Comparator): Provided with proficiency based progression training supported by technology enhanced learning
  Interventions: Behavioral: proficiency based progression training
- Historical controls (No Intervention): no extra training provided

INTERVENTIONS:
Behavioral: proficiency based progression training — proficiency based progression training supported by technology enhanced learning
  Arms: Proficiently Trained interns -

SUMMARY:
Incorrect labelling of blood samples occurs at a rate of 1% in the general laboratories and 6% in Blood Transfusion Laboratories. The most serious error 'Wrong Blood in Tube' (WBIT) occurs when blood is taken from the intended patient, but labelled with another patient's details. Consequences may include, misinterpretation of a patient's diagnosis or clinical status, incorrect referral or treatment of a patient, or in the worst case scenario, incorrect cross matching for blood of the wrong blood group, which may lead to catastrophic outcomes, including death.

The root causes for these errors is failure to identify the patient correctly and failure to correctly label the blood tubes at the bedside. To date, despite significant initiatives, it has proved very difficult to eradicate or reduce the error rate. Our project involves a novel, technology enhanced learning approach using proficiency based progression in a prospective randomised controlled methodology to significantly reduce this error.

This approach to learning is more efficient and effective than the traditional approach of repeated practice and is made possible with metric-based simulations. This project will reduce the incidence of adverse events and avoidable medical errors associated with sampling and labelling errors including WBITs. This will be achieved by training healthcare practitioners to a proficiency standard in venepuncture. Thereby minimising the failure of health care professionals to identify the patient correctly and failure to correctly label the blood tubes at the bedside.

This project's impact will deliver reduced sampling and labelling errors -including WBITs by a factor of 40-69%. Reductions of this magnitude will have profound national and international implications on how these types of skills are acquired and quality assured. This would result in improved patient safety and savings of over €500,000 at Cork University Hospital and if applied nationally result in exchequer savings of millions of euro annually.

DETAILED DESCRIPTION:
The goal of the study is identification, development and operational definition and then validation of phlebotomy performance Metrics which will be used to characterize the optimal performance of healthcare practitioner's execution of phlebotomy. These validated Metrics will serve as an educational and training tool to improve and quality assure phlebotomy training. The validated metrics will be used to produce validated metric-based simulations which will be used to establish a training benchmark based on experienced clinicians' performance. It will also be used to underpin deliberate practice in simulated training.

By introducing proficiency-based progression training supported by technology enhanced learning we aim for reductions in the error rates of wrong blood in tube of 40 to 69%.

Objective 1 To characterize the process of taking a blood sample correctly and the correct process for labelling a blood sample bottle and laboratory request form to reduce the incidence of wrong blood in tube.

This will involve metric development and metric validation of the process of taking a blood sample correctly and the correct process for labelling a blood sample bottle and laboratory request form - as a result of a consultative process, including qualitative analysis of WBIT errors.

Objective 2 To quantitatively define a proficiency benchmark and then to design training to the proficiency standard and assessment of proficiency up to and including real time feedback to the doctor and patient in the clinical arena.

Objective 3 Design a new approach to training including assessment using technology enhanced learning, incorporating online learning and simulation based training of taking a blood sample to a proficiency standard.

Objective 4 To implement the training and assessment in the highest risk groups and document the effectiveness of the intervention.

The training will be delivered to all interns commencing work at Cork University Hospital on July 10th 2017 as proficiency based progression simulation training with additional systematic proximate feedback.

Data from each training group will be identified using the laboratory tracking quality system and using comparison with the historical data from the previous year(s).

Objective 5 To use the research data generated to recommend an evidence based training and competency assessment approach to health care providers in Ireland, together with evidence based individual feedback for any residual errors. This will allow us to internationally address the universal problem of sample mislabeling and WBIT.

ELIGIBILITY:
Inclusion Criteria:

All historical interns blood samples from July to Sept 2016 All interns who receive training and working at Cork University Hospital from July to Sept 2017

Exclusion Criteria:

Interns in 2017 who do not attend for training

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2017-07-05 (Actual); Primary Completion 2018-07-03 (Actual); Study Completion 2018-07-03 (Actual)

PRIMARY OUTCOMES:
WBIT | 3 months
  Wrong blood in tube

SECONDARY OUTCOMES:
wrong bottle type | 3 months
  incorrect bottle type used
under filled samples | 3 months
  number of under filled samples which did not allow analysis
clotted samples | 3 months
  Number of clotted samples
haemolysed samples | 3 months
  number of haemolysed haematology samples
Mislabelling | 3 months
  Mislabelling of forms/bottles in blood bank

CONTACTS AND LOCATIONS:
Overall Officials: Mary Cahill, MD, Study Chair — UCC
Locations (1):
- CUH, Cork, Ireland

IPD SHARING:
Plan to Share IPD: Yes
Available by contacting Principal Investigator
Supporting Information: Study Protocol, ICF, CSR
Time Frame: 6 months
Access Criteria: Determined by principal investigator